CLINICAL TRIAL: NCT05366647
Title: Longterm Comparison of Gonioscopy-assisted Transluminal Trabeculotomy and Canaloplasty in Open-angle Glaucoma Treatment
Brief Title: GATT Versus Canaloplasty (GVC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Joanna Konopińska, Head of Ophthalomogy, Principal Investigator, Clinical Professor, Medical University of Bialystok
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1777
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma, Open-Angle
Keywords: Gonioscopy-assisted Transluminal Trabeculotomy; Canaloplasty; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Canaloplasty (Active Comparator): Canaloplasty ab externo
  Interventions: Procedure: Gonioscopy-assisted Transluminal Trabeculotomy
- Gonioscopy-assisted Transluminal Trabeculotomy (Active Comparator): Gonioscopy-assisted Transluminal Trabeculotomy ab interno
  Interventions: Procedure: canaloplasty

INTERVENTIONS:
Procedure: canaloplasty — canaloplasty ab interno with tensioning suture
  Arms: Gonioscopy-assisted Transluminal Trabeculotomy
Procedure: Gonioscopy-assisted Transluminal Trabeculotomy — Gonioscopy-assisted Transluminal Trabeculotomy ab interno
  Arms: Canaloplasty

SUMMARY:
Study aims to compare the effectiveness and safety profile of Gonioscopy-assisted Transluminal Trabeculotomy and canaloplasty, in order to find out if one operation is superior to the other. Both procedures are performed in patients with medically uncontrolled open-angle glaucoma. Canaloplasty is a recently newly introduced procedure, which showed encouraging results without antimetabolite usage intra- and postoperatively. Gonioscopy-assisted Transluminal Trabeculotomy is the procedure that aims the same mechanism of aqueous outflow, however is perform with ab interno approach, which comprise it to the minimally invasive glaucoma surgery techniques. Purpose of the study is to compare both surgeries concerning success rate, intraocular pressure, medication burden and complications rate. So far there is no comparison of the Gonioscopy-assisted Transluminal Trabeculotomy and canaloplasty available.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older (Adult, Older Adult)
* patients with confirmed uncontrolled open angle glaucoma
* no prior glaucoma surgery (once laser trabeculoplasty or cyclophotocoagulation) allowed

Exclusion Criteria:

* angle closure glaucoma
* congenital glaucoma
* inflammatory glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
success rate (complete and qualified success) | 12 months
  Success is defined: 1. IOP < 21 mmHg and at least 20% IOP change from baseline 2. IOP < 18 mmHg
success rate (complete and qualified success) | 24 months
  Success is defined: 1. IOP < 21 mmHg and at least 20% IOP change from baseline 2. IOP < 18 mmHg

SECONDARY OUTCOMES:
IOP, medication, complications | 12 months
  intraocular pressure change, medication postoperatively, complications intra- and postoperatively
IOP, medication, complications | 24 months
  intraocular pressure change, medication postoperatively, complications intra- and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Konopińska, Principal Investigator — Medical University of Bialystok, Poland
Locations (1):
- Ophthalmology Clinic Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
All materials and information are available upon an e-mail request on principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years